CLINICAL TRIAL: NCT02906306
Title: EFFECTS OF INDIVIDUAL AND GROUP OCCUPATIONAL THERAPY ON GENERAL SELF-EFFICACY AND PSYCHOLOGICAL WELL-BEING IN OLDER ADULTS
Brief Title: Effects of Individual and Group Occupational Therapy on General Self-Efficacy, Psychological Well-Being, Personal Independence and Occupational Therapy in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Abel Toledano-González, Occupational Therapy, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01/2012
Record Dates: First submitted 2016-09-07; First posted 2016-09-20 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Individuality; Self-Efficacy; Well-being
Keywords: Older adults; Occupational Therapy; Self-Efficacy; Psychological Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual Occupational therapy (Experimental): In Individual Occupational Therapy treatment the activities included personal independence training (ADLs), sensory-motor stimulation activities, cognitive stimulation (attention, memory, language and executive function) and animal-assisted therapy (AAT).
  Interventions: Behavioral: Individual Occupational Therapy
- Group Occupational therapy (Experimental): In group Occupational Therapy treatment the activities included personal independence training (ADLs), sensory-motor stimulation activities, cognitive stimulation (attention, memory, language and executive function) and animal-assisted therapy (AAT) and psychosocial skills training.
  Interventions: Behavioral: Group Occupational Therapy

INTERVENTIONS:
Behavioral: Individual Occupational Therapy — 45 minutes 3 times per week 6 months in nursing homes (A and B)
  Arms: Individual Occupational therapy
Behavioral: Group Occupational Therapy — 45 minutes 3 times per week 6 months in nursing homes (A and B)
  Arms: Group Occupational therapy

SUMMARY:
The objective of this study is to determine whether individual and/or group occupational therapy leads to changes in generalized self-efficacy and psychological well-being, and to identify the type of therapy that has the best effects on older adults.

DETAILED DESCRIPTION:
Objective

The main objective of this study is to determine whether individual and/or group occupational therapy leads to changes in generalized self-efficacy and psychological well-being, and to identify the type of therapy that has the best effects on the population of older adults. In addition, the investigators aim to determine whether there is a relationship between the different domains of psychological well-being and the sense of general self-efficacy.

Design

The research draws on a randomized experimental intervention study with a pre-post design. It compares two groups: one receiving individual therapy and the other, group therapy.

Setting

The intervention was conducted at two state-assisted residential care centers for older adults in Málaga (Spain). Each participant was first interviewed to gather sociodemographic data (age, gender, education level) as well as to verify that their scores for cognitive levels and the required skills and capabilities were sufficient to participate in the study. During this interview, the aim and length of the intervention was explained and an invitation to participate was given. All participants gave their informed consent. The care center and the Ethics Committee of the University of Málaga authorized the study. The same cognitive and emotional screening was conducted before and after the intervention. In each care center participants were randomly assigned to the two treatment groups.

Subjects

From an initial sample of 112 residents, a final sample of 74, divided into two groups of 37, was included in the study. For both groups, the inclusion criteria were: 1) able to read; 2) having normal cognitive function, scoring >22 on the Mini Mental Scale Examination, the cut-off point according to the scoring instructions of the adapted version for the Spanish population.

Method

In April 2014, after the sample was selected, participants were randomized to two groups of 34. Following assessment, the intervention began in May. The intervention lasted 6 months, after which participants were re-assessed.

The instruments used were Van Dierendonck's Spanish adaptation of Ryff´s Psychological Well-being Scale, comprising 39 items and with an internal consistency of between 0.78 and 0.81 and the Spanish adaptation of Schwarzer and Jerusalem's General Self-Efficacy Scale (GSE), with an internal consistency of 0.84 (Cronbach's alpha).

Activities were conducted in three 45-minute sessions per week. In both treatment modalities the activities included personal independence training (ADLs), sensory-motor stimulation activities, cognitive stimulation (attention, memory, language and executive function) and animal-assisted therapy (AAT). The group occupational therapy participants also received psychosocial skills training.

To describe the sample, the investigators used descriptive statistics for quantitative and qualitative variables. To analyze differences in the main study variables we applied the t-student test or the Mann-Whitney U test, depending on whether or not they followed a normal distribution. Chi square testing was used to determine the existence of differences in distribution by gender, age and educational level. To analyze the main dependent variables (self-efficacy and well-being) we conducted a repeated measures ANOVA for intra-subject and inter-subject factors. Statistical significance was established at p<0.05. Data were analyzed using SPSS, version 21.0.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read
* Have normal cognitive function scoring >22 on Mini Mental Scale Examination
* Sign informant consent
* Apply the recommendations

Exclusion Criteria:

* Advanced cognitive impairment
* Fear of animals
* Miss three time
* Visual impairment
* Multiple disorders
* Hearing impairment

Ages: 78 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Ryff Questionnaire | 6 months
  The scale of psychological well-being Ryff is formed by the complete version of 39 items with Likert responses it 1-6. The main objective this scale is to measure the degree of psychological well-being of personaa through 6 dimensions: purpose in life, self-acceptance, positive relationships, autonomy, environmental mastery and personal growth
General Self-efficacy | 6 months
  The scale of generalized self-efficacy is a self informed through 10 items with 1-4 Likert scale responses. The main objective is to measure the degree of generalized self-efficacy of the person across 10 assertions with 4 possible answers above, in which the option that best reflects what the person thinks is marked
Barthel Index | 6 months
  Barthel index measured through 10 items the level of dependence of the person performing the activities of daily life can vary between 0 (completely dependent) to 100 (completely independent)
Minimental MMSS | 6 months
  The MMSE is composed of 13 items to assess with scores (0,1,2,3,4,5) according answer. the main objective is to briefly assess the mental state and allow observe the degree of progression of cognitive status through the following areas: orientation, fixation, concentration and calculation, memory, language and construction.
Geriatric Depression Scale (GDS) | 6 MONTHS
  Geriatric Depression Scale consists of 15 items (10 negative and 5 positive) through answers (yes / no) whose content focuses on cognitive behavioral aspects related to special characteristics of the population. The main objective is to facilitate the assessment of depression in the geriatric population.

CONTACTS AND LOCATIONS:
Locations (1):
- Malaga, Málaga, Malaga, Spain

REFERENCES:
- [Derived] Toledano-Gonzalez A, Labajos-Manzanares T, Romero-Ayuso DM. Occupational Therapy, Self-Efficacy, Well-Being in Older Adults Living in Residential Care Facilities: A Randomized Clinical Trial. Front Psychol. 2018 Aug 7;9:1414. doi: 10.3389/fpsyg.2018.01414. eCollection 2018. PMID 30131748